CLINICAL TRIAL: NCT04347915
Title: A Single Blind, Randomized, Placebo-controlled, Multi-center Phase 2 Study to Evaluate the Safety and Efficacy of Clevudine in Patients Diagnosed With Moderate COVID-19
Brief Title: The Phase 2 Study to Evaluate the Safety and Efficacy of Clevudine in Patients With Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BK-CLV-201
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Coronavirus disease-19(COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — clevudine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clevudine (Experimental): Clevudine 120mg (4 capsules) once a day will be administered orally and can be taken regardless of food intake for 14 days (up to 21 days)
  Interventions: Drug: Clevudine
- Placebo (Placebo Comparator): Matching Placebo (4 capsules) once a day will be administered orally and can be taken regardless of food intake for 14 days (up to 21 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clevudine — Clevudine 120mg once a day for 14 days (up to 21 days)
  Arms: Clevudine
Drug: Placebo — Matching Placebo once a day for 14 days (up to 21 days)
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to assess the safety and efficacy of Clevudine 120 mg versus placebo once daily administration with standard of care therapy for 14 days (maximum up to 21 days) in patients with moderate COVID-19.

ELIGIBILITY:
Key Inclusion Criteria:

1. Over 19 years of age
2. COVID-19 confirmed by a real-time RT-PCR tests 4 days prior to clinical trial enrollment
3. Patients with peripheral capillary oxygen saturation (SPO2) greater than 94% at the time of screening
4. Patients whose body temperature is measured according to the measured area without taking a fever reducer during screening:

   [armpit of greater than 37.0 °C or an oral of greater than 37.2 °C; Patients with rectum greater than 37.6 °C or eardrum greater than 37.5 °C] (Notes: Although you take a fever reducer, you can still be enrolled in after investigator's judgement whether there is fever or not.)
5. Patients with evidence of lung invasions as a result of radiation tests

Exclusion Criteria:

1. Patients who need breathing device (for example, Invasive ventilation, Invasive mechanical ventilation, Extra-corporeal membrane oxygenation).
2. Patients who participated in other clinical trials related to COVID-19.
3. Patients who were administered drugs directly to COVID-19 24 hours prior to the start of the study.
4. Patients whose AST or ALT has increased by more than 5 times the normal lab value.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
The rate of subjects tested as negative SARS-Coronavirus-2 (SARS-CoV-2) | within 15days
  The primary efficacy endpoint for this clinical trial is the rate of patients with negative SARS-Coronavirus-2 (SARS-CoV-2) in a two-day continuous Real-Time-RT-PCR test from baseline to before the 15th day.

SECONDARY OUTCOMES:
The rate of subjects tested as negative SARS-Coronavirus-2 (SARS-CoV-2) in consecutive two days of Real-Time RT-PCR tests | Day 4, 8, 11, 15, 22, 29(or EOT) day comparing the baseline
The rate of subjects indicated by the improvement of lung invasive | within Day 29 (or EOT)
The change of viral load | Day 4, 8, 11, 15, 22, and 29(or EOT) comparing the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Woo-Joo Kim, M.D.,Ph.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea